CLINICAL TRIAL: NCT02452112
Title: An Open-Label, Single and Multiple-Dose, Two-Period, Consecutive Study in Healthy Chinese Subjects to Assess the Pharmacokinetic Profiles, Safety and Tolerability of Lidocaine Patch 5%.LIG13-CN-101 Study
Brief Title: Efficacy and Safety of 5% Lidocaine Patch With Placebo Patch in Subjects With Herpes Zoster Associated Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mundipharma (China) Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIG13-CN-301
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Herpes Zoster Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Active Comparator): Active arm with administration of active 5% Lidocaine patch
  Interventions: Drug: 5% Lidocaine patch
- Placebo (Placebo Comparator): Placebo arm with administration of placebo patch
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 5% Lidocaine patch — 5% Lidocaine patch to be placed on the site of pain
  Other Names: Lignopad
  Arms: Lidocaine
Drug: Placebo — Placebo patch to be placed on the site of pain
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study designed to assess the efficacy and safety of 5% lidocaine patch, following placebo or active patch applications in placebo insensitive subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 to 85 years of age.
2. Subjects must have herpes zoster associated pain present for ≥1 months after healing of the acute herpes zoster skin rash and not located on the face, scalp; the diagnosis will be based on physical examination and review of available medical records confirming an episode of herpes zoster.
3. Herpes zoster associated pain must be of at least moderate severity, defined as the average pain level ≥40 mm on a 100 mm visual analog scale (VAS slide ruler)

Exclusion Criteria:

1. Subjects with signs of cord or brainstem injury from herpes zoster.
2. Presence of another pain problem of greater severity than their herpes zoster associated pain.
3. Subjects who have undergone neurolytic nerve blocks or ablative neurosurgical procedures for control of herpes zoster associated pain

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2014-11-02 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Change of VAS score | over 24 hour from baseline to the post-treatment over time during double-blind period
  Mean change in the mean pain VAS score

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Beijing University People's Hospital, Beijing, Beijing Municipality
  - Air force general hospital, Beijing
  - Beijing friendship hospital, Beijing
  - Beijing university first hospital, Beijing
  - Beijing university third hospital, Beijing
  - The first affiliated hospital of Jilin university, Changchun
  - Xiangya hospital central south university, Changsha
  - South West Hospital, Chengdu
  - First affiliated hospital of Chongqing medical university, Chongqing
  - The first affiliated hospital of Dalian university, Dalian
  - Guangzhou general hospital, Guangzhou
  - The first affiliated hospital of Zhejiang university, Hangzhou
  - Shandong dermatology hospital, Jinan
  - The second affiliated hospital of Kunming medical college, Kunming
  - China dermatology research center, Nanjing
  - Shanghai Huashan hospital, Shanghai
  - Shanghai Ruijin Hospital, Shanghai
  - Shengjing Hospital, Shenyang
  - The fourth affiliated hospital of Hebei medical university, Shijiazhuang
  - General hospital of Tianjin medical university, Tianjin
  - Xijing Hospital, Xi'an